CLINICAL TRIAL: NCT07040111
Title: Efficacy and Safety of a 4-Step Versus a 5-Step Egg Ladder in Children With IgE-Mediated Hen's Egg Protein Allergy: Protocol for an Open-Label Randomized Controlled Trial
Brief Title: Efficacy and Safety of Egg Ladders in Children With IgE-Mediated Hen's Egg Protein Allergy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Andrea Horvath-Stolarczyk, Associate Professor, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE2025
Record Dates: First submitted 2025-06-12; First posted 2025-06-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Food Allergy; Egg Allergy; Hen Egg Allergy
Keywords: children; egg ladder; IgE-mediated hen egg allergy
MeSH Terms: conditions — Food Hypersensitivity; Egg Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4-Step Egg Ladder (Experimental)
  Interventions: Other: oral food challenge (OFC)
- 5-Step Egg Ladder (Active Comparator)
  Interventions: Other: oral food challenge (OFC)

INTERVENTIONS:
Other: oral food challenge (OFC) — oral food challenges with subsequent steps of a 4-step egg ladder (muffin [1.5 g of hen's egg protein per portion], pancake, hard-boiled egg, soft-boiled egg)
  Arms: 4-Step Egg Ladder
Other: oral food challenge (OFC) — oral food challenges with subsequent steps of a 5-step egg ladder (muffin [0.75 g of hen's egg protein per portion], muffin [1.5 g of hen's egg protein per portion], pancake, hard-boiled egg, soft-boiled egg)
  Arms: 5-Step Egg Ladder

SUMMARY:
Hen's Egg Allergy is one of the most common food allergies in early childhood. The first-line treatment is the elimination of hen's egg proteins from the child's or maternal diet.

Available data from the literature indicate that most children with hen's egg allergy acquire tolerance to hen's egg proteins with age. An assessment of tolerance acquisition to them is commonly performed using egg ladder. However, scientific evidence regarding the effectiveness and safety of the egg ladder in children with hen's egg allergy is limited. Currently, there is no standardised egg ladder protocol, and different versions of the ladder and recommend by scientific societies in various countries.

This study aims to assess the effectiveness and safety of the 4-step egg ladder (4-EL) compared to the 5-step egg ladder (5-EL) in children with IgE-mediated hen's egg allergy. This is an open-label, randomised superiority trial with two parallel arms and a 1:1 allocation ratio.

DETAILED DESCRIPTION:
Introducing baked egg into the diet of children with hen's egg allergy has been shown to potentially accelerate the development of tolerance to raw egg. However, there is no standardised egg ladder protocol, and different scientific societies across countries recommend varying versions.

This study aims to assess the effectiveness and safety of the 4-step egg ladder (4-EL) compared to the 5-step egg ladder (5-ML) in children with IgE-mediated hen's egg allergy.

An open-label randomised trial with two parallel arms in two departments of the same academic hospital will be performed. A total of 84 children with IgE-mediated hen's egg allergy will be allocated to introduce hen's egg into their diet according to either 4-EL or 5-EL with a 6-week break period between subsequent steps. Oral food challenge (OFCs) with tested products at each subsequent step of the egg ladder will be conducted in hospital settings. The primary outcome is the percentage of children who acquire tolerance to soft-boiled hen's egg (almost raw hen's egg proteins), as determined by a negative OFC at the final step of the EL. Soft-boiled egg will be administered at the end of the observation period (18 or 24 weeks, depending on the assigned study arm). The challenge dose will consist of 0,5-1 egg for children aged 1-3 years and 1 egg for those aged 4-5 years, corresponding to a maximum total of 6 g of hen's egg proteins.

Secondary outcomes will include the percentage of children with a negative OFC to each egg ladder step; the percentage of children with anaphylaxis (both those who were treated and who were not treated with adrenaline); the percentage of children with exacerbation of atopic dermatitis; growth; compliance; and quality of life of the caregivers and parents' anxiety about adverse events during their child's OFC.

The statistical analyses will be conducted with StatsDirect. The Mann-Whitney U test will be used to compare the means of continuous variables if non-normal distribution will be assessed. Proportions will be compared with the Fisher exact test. The difference in study groups was considered significant when the P value will be <05. The results of this study will be analyzed on the basis of intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 months and ≤ 5 years.
* Diagnosis of IgE-mediated HEA confirmed according to the EAACI guidelines by a positive OFC with hen's egg proteins. In children with high-risk HEA (e.g., history of anaphylaxis), diagnosis can be based on elevated specific IgE levels (3.5 kU/l) to hen's egg proteins and/or individual egg components and/or positive skin tests.
* On a therapeutic elimination diet for at least 6 months, measured from the last allergic reaction to egg (in accordance with BSACI guidelines).
* Eligible regardless of the risk of systemic reactions (e.g. anaphylaxis) or asthma.
* Good general health.
* Written informed consent signed by the child's guardians.
* Demonstrated good cooperation from the patient's guardians.

Exclusion Criteria:

* Confirmed wheat allergy and/or celiac disease.
* Uncontrolled asthma, defined as the presence of shortness of breath, cough, chest tightness, or auscultatory changes despite treatment.
* Signs of exacerbation of a chronic disease.
* Signs of acute infectious disease (e.g. acute rhinitis, cough, subfebrile or febrile states).
* Signs of exacerbation of another allergic disease (e.g., conjunctivitis, allergic rhinitis, atopic dermatitis).
* Anaphylaxis due to hen's egg proteins within the last 6 months.
* Use of antihistamines within 3-10 days before the challenge (depending on the drug and indication; time-limited contradiction - relative exclusion criterion).
* Acquired tolerance to baked hen's egg proteins or advancement to a higher step of the egg ladder.
* Use of immunosuppressive drugs or immunotherapy.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the percentage of children who acquire tolerance to soft-boiled hen's egg (almost raw hen's egg proteins) | Soft-boiled egg will be administered at the end of the observation period (18 or 24 weeks, depending on the assigned study arm).
  The primary outcome is the percentage of children who acquire tolerance to soft-boiled hen's egg (almost raw hen's egg proteins), as determined by a negative OFC at the final step of the EL.
  The challenge dose will consist of 0.5-1 egg for children aged 1-3 years and 1 egg for those aged 4-5 years, corresponding to a maximum total of 6 g of hen's egg proteins.

SECONDARY OUTCOMES:
The percentage of children with a negative OFC at each step of the EL protocol upon completion of the study's observation period | 18 weeks and 24 weeks, depending on the study arm
  Calculated as the proportion of children tolerating the full planned dose for each step.
The percentage of children who experienced anaphylaxis | During the observation period (18 or 24 weeks, depending on study arm),
  The proportion of children who experience anaphylaxis defined as reactions with severity grades 3-5 according to the updated 2023 WAO clinical criteria for anaphylaxis.
The proportion of children with anaphylaxis (grades 3-5, per 2023 WAO criteria) who required epinephrine administration. | Measured during the observation period (18 or 24 weeks, depending on the study arm).
  The proportion of children who experienced anaphylaxis and required epinephrine will be reported in three categories:
  * those who require one or two doses of intramuscular epinephrine with a good clinical response (less severe reaction, grade 3),
  * those who require more than 2 doses of intramuscular epinephrine,
  * those with lack of significant clinical improvement after two doses (severe reactions, grades 4-5).
The proportion of children who experienced systemic allergic reactions (SAR) of grades 1, 2, and 3 according to the 2023 WAO grading system. | Measured during the observation period (18 or 24 weeks, depending on the study arm).
  The proportion of children who experienced SAR will be reported in three categories:
  * grade 1: includes nausea and/or mild abdominal pain without altered activity;
  * grade 2: persisting (≥20 mins) and non-distractable abdominal pain and/or vomiting (not due to gag or taste aversion) and/or diarrhea;
  * grade 3: severe, persistent (≥20 minutes), intractable abdominal pain and/or vomiting (excluding retching or taste aversion) and/or diarrhea, assessed during each OFC.
In the subgroup of children with atopic dermatitis, changes in the total score of the oSCORAD index will be assessed. before and after each OFC. | Upon completion of the observation period (18 or 24 weeks, depending on the assigned study arm).
  The maximum score on the oSCORAD scale is 83 points (in the most severe cases, an additional 10 points can be added for changes that disfigure or limit the patient's functioning), the minimum score is 0 points; the more points, the greater intensity of changes. Any documented exacerbation of atopic dermatitis symptoms following OFC will be also recorded.
Change in age-adjusted z-scores for weight and length/height, evaluated using the WHO growth charts. | During the observation period (18 or 24 weeks, depending on study arm).
Change in the total score of the FAQLQ-PF. | At the end of the observation period (18 weeks and 24 weeks, depending on the study arm) from baseline.
  The questionnaire is divided into three domains: emotional impact, food anxiety, and social and dietary limitations. The total score is calculated as the mean of three subscales. The minimum score is 0, the maximum score is 6. The lower the score, the more life affecting the allergy is.
Mean difference in caregiver anxiety levels, measured by the Subjective Units of Distress Scale (SUDS) | Prior to each OFC, between study groups at each time point (18-24 weeks, depending on the study arm).
  parents will rate their level of anxiety on a scale from 1 to 100, where 0 represents no anxiety or complete relaxation, and 100 represents extreme anxiety, the worst ever experienced.
The proportion of children with full adherence to the intervention protocol. | at the end of the observation period (18 or 24 weeks, depending on the assigned study arm)
  The proportion of children with full adherence to the intervention protocol, defined as consumption of at least one portion of a tolerated hen's egg proteins dose three times during last week of break in period, in the same form and quantity as tested during the OFC. Data will be collected through the Egg Ladder Monitoring Diary and assessed throughout each break in period (between the following steps of each ladder).

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Szajewska, MD, Professor, Principal Investigator — Medical University of Warsaw; Anna Nowak-Węgrzyn, MD, Professor, Principal Investigator — Collegium Medicum, University of Warmia and Mazury, Olsztyn, Poland; New York Univeristy, Grossmann School of Medicine; Andrea Horvath, MD, PhD, Principal Investigator — Medical Univeristy of Warsaw; Joanna Jerzyńska, MD, PhD, Principal Investigator — Medical Univeristy of Lodz
Locations (2):
- Poland (2):
  - Medical Univeristy of Warsaw, Department of Paediatrics, Warsaw
  - Medical Univeristy of Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
The results of this RCT, whether positive or negative, will be published in a peer-reviewed journal (data will be submitted to the first journal after 3-6 months from study completion). Abstracts will also be submitted to relevant national and international conferences.
  The datasets used and/or generated during this study will be made available from a given author upon reasonable request, after the publication of results, no later than 3 years from the completion of data analysis.
Supporting Information: Study Protocol
Time Frame: After the publication of results, no later than 3 years from the completion of data analysis with no end date.
Access Criteria: Upon reasonable request.

REFERENCES:
- [Derived] Horvath A, Bujnowska A, Strozyk A, Zemla M, Nowak-Wegrzyn A, Grzela K, Jerzynska J, Szajewska H. Efficacy and safety of a 4-step versus a 5-step egg ladder in children with IgE-mediated hen's egg protein allergy: protocol for an open-label randomized controlled trial. Front Allergy. 2025 Sep 15;6:1658186. doi: 10.3389/falgy.2025.1658186. eCollection 2025. PMID 41031391